CLINICAL TRIAL: NCT03780374
Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2018_37
Record Dates: First submitted 2018-11-30; First posted 2018-12-19 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Each participant will be treated with sound principle 1, 2 and 3 in a crossover design.
Who Masked: Participant
Masking Description: The participant's will not know which intervention will be applied.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sound Processing Principle 1 (Active Comparator): Sound Processing Principle 1 will be applied in the hearing aid.
  Interventions: Device: Phonak Audéo L2M with Sound Processing Principle 1
- Sound Processing Principle 2 (Experimental): Sound Processing Principle 2 will be applied in the hearing aid.
  Interventions: Device: Phonak Audéo L2M with Sound Processing Principle 2
- Sound Processing Principle 3 (Experimental): Sound Processing Principle 3 will be applied in the hearing aid.
  Interventions: Device: Phonak Audéo L2M with Sound Processing Principle 3

INTERVENTIONS:
Device: Phonak Audéo L2M with Sound Processing Principle 1 — Compensation of a hearing loss with Sound Processing Principle 1.
  Arms: Sound Processing Principle 1
Device: Phonak Audéo L2M with Sound Processing Principle 2 — Compensation of a hearing loss with Sound Processing Principle 2.
  Arms: Sound Processing Principle 2
Device: Phonak Audéo L2M with Sound Processing Principle 3 — Compensation of a hearing loss with Sound Processing Principle 3.
  Arms: Sound Processing Principle 3

SUMMARY:
A methodical evaluation of novel sound changing principles in CE-labelled Sonova brand hearing instruments (e.g. Phonak hearing instruments) is intended to be conducted on hearing impaired. These sound changing principles are enabled by respective hearing instrument algorithms. The aim of the study is to investigate and asses strength and weaknesses of these novel sound changing principles in terms of hearing performance to determine their application in hearing instruments (Phase of development). Both, objective laboratory measurements as well as subjective evaluations in real life environment will be carried out. This will be a controlled, single blinded and randomized active comparator clinical evaluation which will be conducted mono-centric at Sonova AG Headquarter based in Staefa.

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years) with and without experience with) hearing aids
* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the medical device in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Speech Intelligibility in Noise | 4 weeks
  The speech intelligibility in noise with the three different sound processing principles will be assessed with the aid of the Oldenburg Sentence Test. The result will be shown in dB (decibel) SRT (Speech Reception Threshold).

SECONDARY OUTCOMES:
Sound Quality - Overall | 16 weeks
  The overall sound quality of sounds with the three different sound processing principles will be assessed with the aid of a questionnaire.
  The results are ratings on a numeric scale, ranging from 0 (bad) to 10 (excellent).
Loudness - Laboratory | 8 weeks
  The loudness of sounds with the three different sound processing principles will be assessed in laboratory with the aid of a MUSHRA (Multi-Stimulus Test with Hidden Reference and Anchor) test.
  The results are ratings on a numeric scale, ranging from 0 (very soft), 50 (just right) to 100 (very loud).
Loudness - Daily Life | 16 weeks
  The loudness of sounds with the three different sound processing principles will be assessed in daily life with the aid of a questionnaire.
  The results are ratings on a numeric scale, ranging from 0 (very soft) to 10 (very loud).
Clarity - Daily Life | 16 weeks
  The clarity of sounds with the three sound processing principles will be assessed with the aid of a questionnaire.
  The results are ratings on a numeric scale, ranging from 0 (very unclear) to 10 (very clear).
Preferred Sound Processing Principle | 16 weeks
  The preferred sound processing principle will be assessed with the aid of a questionnaire.
  The results will be a ranking, ranging from 1 (most preferred) to 3 (least preferred).
Naturalness - Daily Life | 16 weeks
  The sound quality with the three different sound processing principles will be assessed with the aid of a questionnaire.
  The results are ratings on a numeric scale, ranging from 0 (unnatural) to 10 (natural).
Localization - Daily Life | 16 weeks
  The ability to localize sounds with the three different sound processing principles will be assessed with the aid of a questionnaire.
  The results are ratings on a numeric scale, ranging from 0 (not at all locatable) to 10 (very well locatable).
Reverberation - Daily Life | 16 weeks
  The reverberation of sounds with the three different sound processing principles will be assessed with the aid of a questionnaire.
  The results are ratings on a numeric scale, ranging from 0 (not at all reverberant) to 10 (very reverberant).
Satisfaction - Overall in Daily Life | 16 weeks
  The overall satisfaction in daily life with the three different sound processing principles will be assessed with the aid of a questionnaire.
  The results are ratings on a numeric scale, ranging from 0 (very dissatisfied) to 10 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland